CLINICAL TRIAL: NCT06264713
Title: Immersive Virtual REality for Treatment of Unilateral Spatial NEglect Due to Stroke Via Eye-tracking Biofeedback (IRENE Project): a Randomized Controlled Trial
Brief Title: Immersive Virtual REality for Treatment of Unilateral Spatial NEglect Via Eye-tracking Biofeedback
Acronym: IRENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE/2023_041
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-06

CONDITIONS: Neglect, Hemispatial; Stroke
Keywords: Neglect; Stroke; Rehabilitation; Virtual Reality
MeSH Terms: conditions — Perceptual Disorders; Stroke

STUDY DESIGN:
Intervention Model Description: Randomised Clinical Trial
Who Masked: Participant, Investigator
Masking Description: Double blind randomisation. The patients and their families/caregivers are blinded with respect to the group allocation. The assessors are not informed about the group allocation for the entire period of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Immersive Virtual Reality (Experimental): Patients will undergo nine sessions of 20 minutes for three sessions/week, for a total of three weeks of treatment. The training consists of 3 different virtual reality tasks specifically designed for neglect training.
  Interventions: Device: Immersive Virtual Reality
- Sham Immersive Virtual Reality (Active Comparator): Patients will undergo nine sessions of 20 minutes for three sessions/week, for a total of three weeks of treatment. The training consists of 3 different virtual reality tasks specifically designed for neglect training.
  Interventions: Device: Sham Immersive Virtual Reality

INTERVENTIONS:
Device: Immersive Virtual Reality — Patients wear a head-mounted-display and will be immersed in a virtual environment. The stimuli will be provided in the left, center and right visual fields. Eye-tracking biofeedback will be provided about the real-time performance during each exercise.
  Arms: Experimental Immersive Virtual Reality
Device: Sham Immersive Virtual Reality — The patients performed the same protocol of the experimental group, differently to the immersive virtual reality group, from session 2 to session 8 (7 sessions), the stimuli will be provided in the center and right visual fields.
  Arms: Sham Immersive Virtual Reality

SUMMARY:
The purpose of this study is to evaluate the effects of a treatment using virtual reality on the recovery of unilateral spatial neglect. The investigators hypothesize that the experimental group underwent to a protocol of active exercises within the virtual environment will show an improvement in the exploratory functions of the left hemispace, investigated with specific scales and clinical tests.

DETAILED DESCRIPTION:
Cerebral stroke is the second cause of death and the third cause of disability worldwide, and the first cause of disability in the elderly. One of the most commonly encountered neuropsychological disorders following a stroke is the unilateral spatial neglect. The estimated prevalence of unilateral spatial neglect after stroke is 30%, with a difference in prevalence between subjects with right (38%) and left (18%) lesions. unilateral spatial neglect constitutes a limit in the progression of the patient's rehabilitation, slows down functional recovery and increases stress and burden on the caregiver. In recent decades there has therefore been an appeal to the use of new technologies for the treatment of unilateral spatial neglect. Among these, virtual reality allows us to overcome some limitations of traditional interventions (reduced ecological validity) and has the advantage of using an artificial environment in the virtual space which allows the execution of tasks that simulate the activities of common life. Furthermore, virtual reality systems offer the opportunity to recreate safe, ecological and personalized 3D environments in which patients must perform specific and controlled actions to achieve a goal. Numerous studies have investigated the effectiveness of training with virtual reality showing that it can improve spatial attention in subjects with unilateral spatial neglect and promote the integration of this ability into daily life activities. To date, the studies available in the literature show that through virtual reality treatment it is possible to find significant improvements in the deficit of unilateral spatial neglect.

Specifically, patients undergoing virtual reality training showed an increase in visual perception of the left hemispace and in head movements on the affected side following virtual reality training compared to controls, maintaining the results at the 3-month follow-up. Although encouraging, the data available to date are the result of clinical studies characterized by high heterogeneity, medium methodological value and small sample size. Further investigations are needed to generalize the results. Within virtual environments, performance is measured objectively and the level of difficulty can be adjusted to gradually increase the complexity of the tasks by reducing the support and feedback provided by the therapist. Furthermore, through the immersive virtual reality it is possible to record all the data regarding the actions carried out by the patient within the virtual scenario and this can be used to create performance indices with which to measure, in a quantitative and objective manner, the progress during the rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

* Ischaemic or hemorrhagic lesion in one hemisphere only (right or left hemiplegia/hemiparesis)
* Presence of unilateral spatial neglect confirmed by neuropsychological examination
* Mini Mental State Examination > 23
* The patient must be able to maintain a sitting position and rotate his head
* Onset acute event no later than 180 days from the date of enrollment

Exclusion Criteria:

* Multiple or bilateral lesions
* Presence of visual difficulties
* Right neglect with associated aphasic deficit (in comprehension)
* Mini Mental State Examination < 23
* Presence of degenerative pathologies, tumors, or other comorbid pathologies
* Epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the Behavioural Inattention Test | Baseline, 4 weeks from baseline, 8 weeks from baseline
  The Behavioural Inattention Test (BIT) allows for the assessment of the presence and extent of unilateral spatial neglect through a series of tests comprising "conventional" subtests (paper and pencil tasks) and "behavioural" subtests that reflect aspects of neglect interference during the performance of daily activities. The results of the BIT provide a detailed overview of the presentation of patients with neglect across a wide range of visuo-spatial tasks. The total score resulting from performance on the conventional subtests is considered pathological if it is below the threshold value of 129 (129/146), with lower scores indicating an increased level of impairment.

SECONDARY OUTCOMES:
Changes in the Copying drawings with or without programming elements | Baseline, 4 weeks from baseline, 8 weeks from baseline
  The drawing copy test with or without programming elements is used to assess constructive praxis. It comprises three items that the subject must copy freehand or with the assistance of some graphic elements of the model already present on the sheet on which they are copying. The scoring is differentiated: for freehand copying, the range is 0-12, while for copying with programming elements, the range is 0-70. In both cases, lower scores indicate an increased impairment of the function.
Changes in the Barrage Test | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Albert's Test is employed to detect the presence of unilateral spatial neglect in stroke patients. In this test, patients are required to cross out all the lines arranged in random orientations on a sheet of paper (A3 format). The score is determined by the number of segments correctly crossed out, for both the right (10 stimuli) and left (11 stimuli) sides. A difference of 1 omission between the right and left sides is considered pathological.
Changes in the Wundt Justrow area illusion test | Baseline, 4 weeks from baseline, 8 weeks from baseline
  The Wundt-Jastrow Illusion Test is utilized to assess the presence of unilateral spatial neglect. It employs the Wundt-Jastrow illusion: two sectors of a circle, equal in shape and size, are perceived as different if they are juxtaposed in a way that one of them appears longer. This phenomenon is consistent for all normal subjects but may disappear in the case of neglect. The subject is presented with 40 boards (A3 format), each containing two stimuli, varied in dimensions, convexity orientation (upward or downward), and the position (right or left) of the misaligned margins that induce the illusion. A score is obtained for "expected" responses and one for "unexpected" responses, depending on whether the critical part of the stimulus is on the right or left. A difference greater than 2 between the number of unexpected responses on the right and left indicates neglect.
Changes in the Kessler Foundation Neglect Assessment Process | Baseline, 4 weeks from baseline, 8 weeks from baseline
  The Kessler Foundation Neglect Assessment Process (KF-NAP™) is used to assess symptoms of spatial neglect in activities of daily living and to assist predicting functional outcomes after a brain damage, such as stroke or traumatic brain injury, in the context of comprehensive clinical evaluation. In addition to the clinical purpose, the KF-NAP™ can be used as an outcome measure in research studies. Behaviours observed in the KF-NAP™ are related to spatial locations in the personal space , the peri-personal space , the extra-personal space, and the mental space. Total scores range from 0 - 30 with higher scores indicating increased disability.
Changes in the Stroke Specific Quality of Life Scale | Baseline, 4 weeks from baseline, 8 weeks from baseline
  The Stroke Specific Quality of Life Scale (SSQoL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke. Total scores range from 49-245 with higher scores indicate better functioning
Changes in the Fugl-Meyer Assessment scale | Baseline, 4 weeks from baseline, 8 weeks from baseline
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment scale. It is designed to assess motor functioning, sensation, balance, joint range of motion and joint pain in patients with post-stroke hemiplegia. Motor score: ranges from 0 (hemiplegia) to 100 points (normal motor performance). Divided into 66 points for upper extremity and 34 points for the lower extremity. Sensation: ranges from 0 to 24 points. Divided into 8 points for light touch and 16 points for position sense. Balance: ranges from 0 to 14 points. Divided into 6 points for sitting and 8 points for standing. Joint range of motion: ranges from 0 to 44 points. Joint pain: ranges from 0 to 44 points. It determine disease severity, describe motor recovery, and to plan and assess treatment. a score range between 96-99 indicates slight motor discoordination; a score between 85 and 95 indicates hemiparesis; and a score ≤ 84 indicates hemiplegia.
Changes in reaction time e time of fixation | Baseline, 4 weeks from baseline, 8 weeks from baseline
  The fixation time expressed in percentage and reaction time expressed in millisecond will be recorded via eye-tracking.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Santa Lucia Foundation, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Esposito E, Shekhtman G, Chen P. Prevalence of spatial neglect post-stroke: A systematic review. Ann Phys Rehabil Med. 2021 Sep;64(5):101459. doi: 10.1016/j.rehab.2020.10.010. Epub 2021 Sep 24. PMID 33246185
- [Result] Navarro MD, Llorens R, Noe E, Ferri J, Alcaniz M. Validation of a low-cost virtual reality system for training street-crossing. A comparative study in healthy, neglected and non-neglected stroke individuals. Neuropsychol Rehabil. 2013;23(4):597-618. doi: 10.1080/09602011.2013.806269. Epub 2013 Jun 14. PMID 23767963
- [Result] De Luca R, Lo Buono V, Leo A, Russo M, Aragona B, Leonardi S, Buda A, Naro A, Calabro RS. Use of virtual reality in improving poststroke neglect: Promising neuropsychological and neurophysiological findings from a case study. Appl Neuropsychol Adult. 2019 Jan-Feb;26(1):96-100. doi: 10.1080/23279095.2017.1363040. Epub 2017 Sep 22. PMID 28937807
- [Result] Yasuda K, Kato R, Sabu R, Kawaguchi S, Iwata H. Development and proof of concept of an immersive virtual reality system to evaluate near and far space neglect in individuals after stroke: A brief report. NeuroRehabilitation. 2020;46(4):595-601. doi: 10.3233/NRE-203014. PMID 32508332
- [Result] Choi HS, Shin WS, Bang DH. Application of digital practice to improve head movement, visual perception and activities of daily living for subacute stroke patients with unilateral spatial neglect: Preliminary results of a single-blinded, randomized controlled trial. Medicine (Baltimore). 2021 Feb 12;100(6):e24637. doi: 10.1097/MD.0000000000024637. PMID 33578583
- [Result] Heyse J, Carlier S, Verhelst E, Vander Linden C, De Backere F, De Turck F. From Patient to Musician: A Multi-Sensory Virtual Reality Rehabilitation Tool for Spatial Neglect. Applied Sciences. 2022; 12(3):1242. https://doi.org/10.3390/app12031242
- [Result] Smith J, Hebert D, Reid D. Exploring the effects of virtual reality on unilateral neglect caused by stroke: Four case studies. Technol. Disabil. 2007;19:29-40. doi: 10.3233/TAD-2007-19104.
- [Result] Kim J, Kim K, Kim DY, Chang WH, Park CI, Ohn SH, Han K, Ku J, Nam SW, Kim IY, Kim SI. Virtual environment training system for rehabilitation of stroke patients with unilateral neglect: crossing the virtual street. Cyberpsychol Behav. 2007 Feb;10(1):7-15. doi: 10.1089/cpb.2006.9998. PMID 17305443
- [Result] Ogourtsova T, Souza Silva W, Archambault PS, Lamontagne A. Virtual reality treatment and assessments for post-stroke unilateral spatial neglect: A systematic literature review. Neuropsychol Rehabil. 2017 Apr;27(3):409-454. doi: 10.1080/09602011.2015.1113187. Epub 2015 Dec 1. PMID 26620135
- [Result] Martino Cinnera A, Bisirri A, Chioccia I, Leone E, Ciancarelli I, Iosa M, Morone G, Verna V. Exploring the Potential of Immersive Virtual Reality in the Treatment of Unilateral Spatial Neglect Due to Stroke: A Comprehensive Systematic Review. Brain Sci. 2022 Nov 20;12(11):1589. doi: 10.3390/brainsci12111589. PMID 36421913
- [Result] Katz N, Ring H, Naveh Y, Kizony R, Feintuch U, Weiss PL. Interactive virtual environment training for safe street crossing of right hemisphere stroke patients with unilateral spatial neglect. Disabil Rehabil. 2005 Oct 30;27(20):1235-43. doi: 10.1080/09638280500076079. PMID 16298925
- [Result] Pedroli E, Serino S, Cipresso P, Pallavicini F, Riva G. Assessment and rehabilitation of neglect using virtual reality: a systematic review. Front Behav Neurosci. 2015 Aug 25;9:226. doi: 10.3389/fnbeh.2015.00226. eCollection 2015. PMID 26379519